CLINICAL TRIAL: NCT01795443
Title: Lumbar Proprioception in Lower Back Pain Patients Versus Healthy Subjects : a Comparative Study on the Effects of Low- and High-frequency Muscle Vibrations
Acronym: Vibrioception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: LOCAL/2012/AD-03; 2012-A01733-40 (Other: RCB number)
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Back Pain
Keywords: vibration; proprioception
MeSH Terms: conditions — Back Pain | interventions — Calibration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (12):
- Healthy volunteers 1 (Active Comparator): The patients in this arm of the study are healthy volunteers with no history of back pain in the last five years (see inclusion/exclusion criteria).
  Propioception measures will be carried out in the following order:
  Intervention: Calibration; Intervention: Practice; Intervention: Measures - no vibration; Intervention: Measures - high vibration; Intervention: Measures - low vibration;
  Interventions: Other: Calibration; Other: Practice; Other: Measures - no vibration; Other: Measures - low vibration; Other: Measures - high vibration
- Healthy volunteers 2 (Active Comparator): The patients in this arm of the study are healthy volunteers with no history of back pain in the last five years (see inclusion/exclusion criteria).
  Propioception measures will be carried out in the following order:
  Intervention: Calibration; Intervention: Practice; Intervention: Measures - no vibration; Intervention: Measures - low vibration; Intervention: Measures - high vibration;
  Interventions: Other: Calibration; Other: Practice; Other: Measures - no vibration; Other: Measures - low vibration; Other: Measures - high vibration
- Healthy volunteers 3 (Active Comparator): The patients in this arm of the study are healthy volunteers with no history of back pain in the last five years (see inclusion/exclusion criteria).
  Propioception measures will be carried out in the following order:
  Intervention: Calibration; Intervention: Practice; Intervention: Measures - high vibration; Intervention: Measures - no vibration; Intervention: Measures - low vibration;
  Interventions: Other: Calibration; Other: Practice; Other: Measures - no vibration; Other: Measures - low vibration; Other: Measures - high vibration
- Healthy volunteers 4 (Active Comparator): The patients in this arm of the study are healthy volunteers with no history of back pain in the last five years (see inclusion/exclusion criteria).
  Propioception measures will be carried out in the following order:
  Intervention: Calibration; Intervention: Practice; Intervention: Measures - high vibration; Intervention: Measures - low vibration; Intervention: Measures - no vibration;
  Interventions: Other: Calibration; Other: Practice; Other: Measures - no vibration; Other: Measures - low vibration; Other: Measures - high vibration
- Healthy volunteers 5 (Active Comparator): The patients in this arm of the study are healthy volunteers with no history of back pain in the last five years (see inclusion/exclusion criteria).
  Propioception measures will be carried out in the following order:
  Intervention: Calibration; Intervention: Practice; Intervention: Measures - low vibration; Intervention: Measures - no vibration; Intervention: Measures - high vibration;
  Interventions: Other: Calibration; Other: Practice; Other: Measures - no vibration; Other: Measures - low vibration; Other: Measures - high vibration
- Healthy volunteers 6 (Active Comparator): The patients in this arm of the study are healthy volunteers with no history of back pain in the last five years (see inclusion/exclusion criteria).
  Propioception measures will be carried out in the following order:
  Intervention: Calibration; Intervention: Practice; Intervention: Measures - low vibration; Intervention: Measures - high vibration; Intervention: Measures - no vibration;
  Interventions: Other: Calibration; Other: Practice; Other: Measures - no vibration; Other: Measures - low vibration; Other: Measures - high vibration
- Back pain patients 1 (Experimental): The patients included in this arm have had back pain for at least 6 months; the origin of this back pain can not be from a previous surgery (see inclusion and exclusion criteria).
  Propioception measures will be carried out in the following order:
  Intervention: Calibration; Intervention: Practice; Intervention: Measures - no vibration; Intervention: Measures - high vibration; Intervention: Measures - low vibration;
  Interventions: Other: Calibration; Other: Practice; Other: Measures - no vibration; Other: Measures - low vibration; Other: Measures - high vibration
- Back pain patients 2 (Experimental): The patients included in this arm have had back pain for at least 6 months; the origin of this back pain can not be from a previous surgery (see inclusion and exclusion criteria).
  Propioception measures will be carried out in the following order:
  Intervention: Calibration; Intervention: Practice; Intervention: Measures - no vibration; Intervention: Measures - low vibration; Intervention: Measures - high vibration;
  Interventions: Other: Calibration; Other: Practice; Other: Measures - no vibration; Other: Measures - low vibration; Other: Measures - high vibration
- Back pain patients 3 (Experimental): The patients included in this arm have had back pain for at least 6 months; the origin of this back pain can not be from a previous surgery (see inclusion and exclusion criteria).
  Propioception measures will be carried out in the following order:
  Intervention: Calibration; Intervention: Practice; Intervention: Measures - high vibration; Intervention: Measures - no vibration; Intervention: Measures - low vibration;
  Interventions: Other: Calibration; Other: Practice; Other: Measures - no vibration; Other: Measures - low vibration; Other: Measures - high vibration
- Back pain patients 4 (Experimental): The patients included in this arm have had back pain for at least 6 months; the origin of this back pain can not be from a previous surgery (see inclusion and exclusion criteria).
  Propioception measures will be carried out in the following order:
  Intervention: Calibration; Intervention: Practice; Intervention: Measures - high vibration; Intervention: Measures - low vibration; Intervention: Measures - no vibration;
  Interventions: Other: Calibration; Other: Practice; Other: Measures - no vibration; Other: Measures - low vibration; Other: Measures - high vibration
- Back pain patients 5 (Experimental): The patients included in this arm have had back pain for at least 6 months; the origin of this back pain can not be from a previous surgery (see inclusion and exclusion criteria).
  Propioception measures will be carried out in the following order:
  Intervention: Calibration; Intervention: Practice; Intervention: Measures - low vibration; Intervention: Measures - no vibration; Intervention: Measures - high vibration;
  Interventions: Other: Calibration; Other: Practice; Other: Measures - no vibration; Other: Measures - low vibration; Other: Measures - high vibration
- Back pain patients 6 (Experimental): The patients included in this arm have had back pain for at least 6 months; the origin of this back pain can not be from a previous surgery (see inclusion and exclusion criteria).
  Propioception measures will be carried out in the following order:
  Intervention: Calibration; Intervention: Practice; Intervention: Measures - low vibration; Intervention: Measures - high vibration; Intervention: Measures - no vibration;
  Interventions: Other: Calibration; Other: Practice; Other: Measures - no vibration; Other: Measures - low vibration; Other: Measures - high vibration

INTERVENTIONS:
Other: Calibration — Subjects will be seated on a table, feet dangling, blindfolded, arms crossed over the chest and held in place by bandages to minimize the visual and proprioceptive inputs that may contribute to the realization of the task.
  The investigator uses an electronic goniometer to measure the maximal extension and flexion during a pelvic pivot. These measures will be used to determine a "target" position midway along the pelvic movement range.
Other: Practice — Propioception test: The movement required is flexion - extension of the lumbar spine without moving the shoulders; it is a pelvic rocking motion. The patients will be helped to the target position by the investigator. After keeping the target position for 5 seconds, they will be asked to completely pivot the pelvis to a forward position, then return to the target position.
  Each subject will have three (non-measured) tries at the proprioception test without vibration, then three tries with low frequency vibration (20 Hertz), and then three tries with high frequency vibration (60 Hertz). Between each series of tries, a 2-minute rest period with walking is required.
Other: Measures - no vibration — The movements required are performed without vibration.
  The movement required is flexion - extension of the lumbar spine without moving the shoulders; it is a pelvic rocking motion. The patients will be helped to the target position by the investigator. After keeping the target position for 5 seconds, they will be asked to completely pivot the pelvis to a forward position, then return to the target position. This test is repeated five times.
  The investigator measures the lumbar angle using an electronic goniometer twice during each of the five tests: once after the patient is helped to the target angle, and once after the patient tries to "remember" the target angle by his/herself.
Other: Measures - low vibration — The movements required are performed with low frequency vibration (20 Hertz on following device: VIBRALGIC 5; manufacturer = Electronique Conseil).
  The movement required is flexion - extension of the lumbar spine without moving the shoulders; it is a pelvic rocking motion. The patients will be helped to the target position by the investigator. After keeping the target position for 5 seconds, they will be asked to completely pivot the pelvis to a forward position, then return to the target position. This test is repeated five times.
  The investigator measures the lumbar angle using an electronic goniometer twice during each of the five tests: once after the patient is helped to the target angle, and once after the patient tries to "remember" the target angle by his/herself.
Other: Measures - high vibration — The movements required are performed with low frequency vibration (20 Hertz on following device: VIBRALGIC 5; manufacturer = Electronique Conseil).
  The movement required is flexion - extension of the lumbar spine without moving the shoulders; it is a pelvic rocking motion. The patients will be helped to the target position by the investigator. After keeping the target position for 5 seconds, they will be asked to completely pivot the pelvis to a forward position, then return to the target position. This test is repeated five times.
  The investigator measures the lumbar angle using an electronic goniometer twice during each of the five tests: once after the patient is helped to the target angle, and once after the patient tries to "remember" the target angle by his/herself.

SUMMARY:
The primary objective of this study is to compare the lumbar proprioception of patients with chronic back pain to that of healthy volunteers during low- and high-frequency muscle vibration.

The order of measures (low frequency of vibration, high frequency vibration and no vibration) is randomized in a cross-over design.

Patients and volunteers are matched by age and body mass index.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

A-Measure the effect of low- and high-frequency vibrations on lumbar repositioning in patients with chronic lower back pain.

B-Measure the effect of low- and high-frequency vibrations on lumbar repositioning in healthy volunteers.

Our working hypothesis is that low frequency vibrations induce an illusion of shortening, and high frequency vibrations induce an illusion of elongation. The variability of the error should not increase.

ELIGIBILITY:
Inclusion Criteria for patients:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient has had chronic low back pain (which did NOT originate in a postoperative setting) for at least 6 months

Inclusion Criteria for healthy volunteers:

* The subject must have given his/her informed and signed consent
* The subject must be insured or beneficiary of a health insurance plan

Exclusion Criteria for patients:

* The patient is under judicial protection, or any kind of guardianship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* The patient has a history of spinal surgery
* The patient has a history of preexisting postural disorder preceding low back pain
* The patient has been treated in the last month (e.g. back pain injections)
* The patient has a balance disorder, blindness, inability to perform the experimental protocol

Exclusion Criteria for healthy volunteers:

* The subject is under judicial protection, or any kind of guardianship
* The subject refuses to sign the consent
* It is impossible to correctly inform the subject
* The subject is pregnant, parturient, or breastfeeding
* The subject has a history of spinal surgery
* The subject has a history of preexisting postural disorder preceding low back pain
* The subject has been treated in the last month (e.g. back pain injections)
* The subject has a balance disorder, blindness, inability to perform the experimental protocol
* The subject has a history of acute low back pain > 15 days or which has resulted in leave from work for more than 7 days in the 5 years preceding the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Measurement erreur | Baseline (day O)
  Measures are made with an electronic goniometer.
  Measurement erreur = (Lumbar angle in the target position) - (lumbar angle in patient-perceived target position)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Dupeyron, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, Gard, France